CLINICAL TRIAL: NCT00242034
Title: Investigation of Cervix Tumor Oxygenation and Microvasculature Using Magnetic Resonance Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00-0152-C
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-08

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Spectroscopy; Contrast Media

INTERVENTIONS:
Procedure: CT and MRI with contrast

SUMMARY:
In cervix cancer tumor oxygen levels and fluid pressure in the tumor have been shown to be related to patient outcome. Analysis of the way tumors enhance after intravenous contrast injection using MRI and CT can be used to determine parameters that relate to tumor blood vessels. In this study we hope to determine if there is a relationship between the enhancement of cervix cancer on MRI and CT and tumor oxygen levels and interstitial fluid pressure. If such a relationship exists then it could help improve the care of patients wiht cervix cancer by allowing for more aggressive therapy of patients with cancer that have more ominous imaging characteristics

DETAILED DESCRIPTION:
MRI is already used routinely in the radiation planning and staging of carcinoma of the cervix. Prognostic factors such as T-stage (local extent), tumor size and lymphadenopathy are routinely obtained from MRI, however some prognostic parameters can only be obtained invasively. Tumor oxygenation correlates with prognosis and response to treatment in patients undergoing radiotherapy for carcinoma of the cervix. Interstitial fluid pressure (IFP) has been shown to correlate with tumor oxygenation as well. Currently the only way to measure these parameters is by using an invasive technique which involves the placement of probes into the tumor and obtaining multiple measurements.

Recent studies have shown that a specific MRI pulse sequences may be able to measure the oxygenation in the microcirculation. A second way of assessing the tumor microvasculature and perfusion is based on the behavior of intravenous contrast agents routinely used in the MRI examination. Estimates of blood volume, and capillary permeability can be made by mathematically modeling the kinetics of an MRI contrast agent. Similar measurements can be performed with CT.

A total of 60 patients will be investigated. Additional images will be obtained from these patients after their routine MRI examination. One set of images is designed to measure a parameter that correlates with tumor oxygen levels. The second set of images will be obtained after the injection of intravenous contrast agent. Using mathematical models a number of parameters will be extracted and correlated with IFP and tumor oxygen measurements.

ELIGIBILITY:
Inclusion Criteria:

* Cervix cancer intended for radiation therapy

Exclusion Criteria:

* Contraindication to contrast enhanced MRI and CT
* Prior therapy for cervix cancer
* Prior pelvic radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Masoom Haider, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret HOspital, Toronto, Ontario, Canada